CLINICAL TRIAL: NCT00899015
Title: Sample Analysis for Terminated Protocol 00-C-0070, Pediatric Phase I Trial of Arsenic Trioxide
Brief Title: Assessing Arsenic Trioxide in Young Patients With Leukemia or Lymphoma Who Were Treated on Clinical Trial NCI-00-C-0070J
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Other Study IDs: 999907221; 07-C-N221; CDR0000570658
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Leukemia; Lymphoma
Keywords: recurrent childhood acute myeloid leukemia; childhood acute promyelocytic leukemia (M3); recurrent childhood acute lymphoblastic leukemia; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent/refractory childhood Hodgkin lymphoma; childhood chronic myelogenous leukemia; atypical chronic myeloid leukemia, BCR-ABL1 negative
MeSH Terms: conditions — Leukemia; Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Burkitt Lymphoma; Recurrence; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative

INTERVENTIONS:
Other: pharmacological study

SUMMARY:
RATIONALE: Studying bone marrow and blood samples from patients with leukemia or lymphoma treated with arsenic trioxide may help doctors learn more about cancer.

PURPOSE: This research study is assessing arsenic trioxide in young patients with recurrent or refractory leukemia or lymphoma who were treated on clinical trial NCI-00-C-0070J.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the pharmacokinetic and pharmacodynamic profiles of arsenic trioxide in pediatric patients treated on protocol NCI-00-C-0070J.

OUTLINE: Bone marrow or peripheral blood mononuclear cells collected during treatment on NCI-00-C-0070J are assessed for pharmacodynamics studies. Plasma cells collected during treatment are assessed for pharmacokinetics studies. Total arsenic (As), inorganic As forms (AsIII and AsV), and methylated metabolites of As are assessed.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed leukemia or lymphoma refractory to standard curative treatment regimens

  * No meningeal leukemia or lymphoma
  * No HIV-related lymphoma
  * No lymphoproliferative diseases
* Received treatment on protocol NCI-00-C-0070J
* Bone marrow or peripheral blood and serum samples collected during treatment on NCI-00-C-0070J are available

PATIENT CHARACTERISTICS:

* See NCI-00-C-0070J

PRIOR CONCURRENT THERAPY:

* See NCI-00-C-0070J

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Estimated)
Dates: Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK)
Pharmacodynamics (PD)
Correlation of PK and PD with clinical parameters, such as age, gender, and dose

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Fox, MD, Principal Investigator — National Cancer Institute (NCI)